CLINICAL TRIAL: NCT01866982
Title: The PREMOD Trial: A Randomized Controlled Trial of Umbilical Cord Milking vs. Delayed Cord Clamping in Premature Infants
Acronym: PREMOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PREMOD; R03HD072934-01 (NIH)
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Intraventricular Hemorrhage
Keywords: umbilical cord milking; delayed cord clamping
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Umbilical Cord Milking (Active Comparator): Milking the umbilical cord 4 times towards the infants at a speed of 20cm/2 seconds
  Interventions: Procedure: Umbilical Cord Milking
- Delayed Cord Clamping (Active Comparator): Delayed clamping of the umbilical cord for 45-60 seconds
  Interventions: Procedure: Delayed Cord Clamping

INTERVENTIONS:
Procedure: Umbilical Cord Milking — Umbilical cord milked toward the neonate four times at a speed of 20cm/2seconds, prior to clamping and cutting umbilical cord. Procedure takes about 10-20 seconds.
  Arms: Umbilical Cord Milking
Procedure: Delayed Cord Clamping — Performed by positioning the baby 20 cm below the placenta for 45-60 seconds prior to umbilical cord clamping and cutting.
  Arms: Delayed Cord Clamping

SUMMARY:
Premature babies can be very sick and have bleeding in the brain. Giving babies more blood before cutting the umbilical cord by delayed cord clamping or umbilical cord milking has been shown to reduce the risk of bleeding in the brain. This may be related to improving perfusion to the brain. However, some studies suggest that delayed cord clamping may not increase hemoglobin or blood volume in babies delivered by cesarean section. Milking the umbilical cord may give more blood in babies delivered by Cesarean Section may improve perfusion and reduce bleeding in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Singleton or multiples pregnancies in patients admitted for medically indicated delivery or in advanced spontaneous preterm labor with imminent delivery at 23 0/7 - 31 6/7 weeks gestation

Exclusion Criteria:

* Planned vaginal breech delivery
* Major fetal abnormalities (defined as those that are lethal or require prenatal or postnatal surgery)
* Fetal death in utero
* Red cell isoimmunization
* Patients who are incapable of informed consent (unconscious, severely ill, mentally handicapped), or are unwilling to undergo randomization
* Placenta accreta or abruption

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Superior Vena Cava Flow | <12 hours of life

SECONDARY OUTCOMES:
Delivery Room Interventions | 10 minutes of life
Hemoglobin | <1 hour
Hemoglobin | 12 hours
Hemoglobin | 4 weeks of life
Neurodevelopmental impairment 18-36 months | 18-36 months
Severe intraventricular hemorrhage (grade 3 or 4) | up to 24 weeks after birth
Phototherapy | up to 24 weeks after birth
  Requirement and length of phototherapy
Ionotropic support | up to 24 weeks after birth
  Requirement and length of ionotropic support
Neonatal intensive care unit (NICU) length of stay | up to 24 weeks after birth
Necrotizing enterocolitis | up to 24 weeks after birth
Number of blood transfusions while in the neonatal intensive care unit | up to 24 weeks after birth
Ventilator time | up to 24 weeks after birth
Apgar score <7 at 5 minutes | at 5 minutes after birth
Umbilical cord pH < 7.0 | up to 30 minutes after birth
Blood pressure in first 2 hours of admission to neonatal intensive care unit | 2 hours after birth
Polycythemia | up to 24 hours of life
Neonatal death | up to 24 weeks of life
Use of uterotonic agents | up to 1 hour after birth
Peak transcutaneous and/or serum bilirubin concentrations | up to 24 weeks after birt
Maternal hemoglobin | within 48 hours after delivery
Intraventricular Hemorrhage detected on Head Ultrasound | up to 24 weeks after birth

OTHER OUTCOMES:
Days on Oxygen | during hospitalization
Vaginal Delivered infants (no difference in interventions) | up to 24 weeks after birth
Cerebral Tissue Oxygenation | Up to 24 hours of life
Cardiac output by electric cardiometry | up to 24 hours of life
Stroke volume by electric cardiometry | Up to 24 hours of life

CONTACTS AND LOCATIONS:
Overall Officials: Anup C Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (3):
- United States (3):
  - Loma Linda Medical Center, Loma Linda, California
  - Sharp Mary Birch, San Diego, California
  - University of California, San Diego, San Diego, California

REFERENCES:
- [Background] Katheria AC, Truong G, Cousins L, Oshiro B, Finer NN. Umbilical Cord Milking Versus Delayed Cord Clamping in Preterm Infants. Pediatrics. 2015 Jul;136(1):61-9. doi: 10.1542/peds.2015-0368. PMID 26122803
- [Background] Katheria A, Garey D, Truong G, Akshoomoff N, Steen J, Maldonado M, Poeltler D, Harbert MJ, Vaucher YE, Finer N. A Randomized Clinical Trial of Umbilical Cord Milking vs Delayed Cord Clamping in Preterm Infants: Neurodevelopmental Outcomes at 22-26 Months of Corrected Age. J Pediatr. 2018 Mar;194:76-80. doi: 10.1016/j.jpeds.2017.10.037. Epub 2017 Dec 12. PMID 29246467